CLINICAL TRIAL: NCT01027143
Title: Obesity & Asthma: Nutrigenetic Response to Omega-3 Fatty Acids
Brief Title: Obesity and Asthma: Nutrigenetic Response to Omega-3 Fatty Acids
Acronym: NOOA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCCJELK23
Record Dates: First submitted 2009-12-03; First posted 2009-12-07 (Estimated); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2016-03

CONDITIONS: Asthma; Obesity
Keywords: Asthma; Obesity; Pharmacogenetics; Nutrigenetics
MeSH Terms: conditions — Asthma; Obesity | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- omega-3 fatty acids (Experimental): 3 softgels (EPA, DHA) twice daily
  Interventions: Dietary Supplement: omega-3 polyunsaturated fatty acids
- control (Placebo Comparator): Soybean oil: 3 matched softgel caps twice daily
  Interventions: Drug: Omega-3 Fatty Acid

INTERVENTIONS:
Dietary Supplement: omega-3 polyunsaturated fatty acids — ProEPA Xtra 1000mg softgels: 3 softgels twice daily
  Other Names: ProEPA Xtra 1000mg softgels
  Arms: omega-3 fatty acids
Drug: Omega-3 Fatty Acid — Soybean oil: 3(age 12-25) matched softgel caps twice daily
  Other Names: Placebo Soybean oil 1000mg soft gels
  Arms: control

SUMMARY:
This project will assess the effectiveness of omega-3 fatty acid supplementation in controlling asthma symptoms among obese asthmatics, and will assess if a person's genes influence response to treatment (personalized medicine). This project may improve our ability to treat asthma and our understanding of the link between obesity and asthma.

DETAILED DESCRIPTION:
Obesity increases the risk for asthma diagnosis in children and adults. With obesity on the rise, a better understanding of this association may become critically important to public health. We will determine the impact of fish oil-derived Eicosapentaenoic acid (EPA) and Docosahexaenoic acid (DHA) on asthma control among obese asthmatics. These omega-3 fatty acids have been shown to: reduce inflammation important to asthma and improve asthma outcomes in an inconsistent manner across previous smaller studies - results that are consistent with a pharmacogenetic influence. There exists evidence that omega-3 fatty acid response displays a pharmacogenetic response related to ALOX5 genotype. Preliminary data suggests that obese individuals are at greater risk for possessing this same ALOX5 variant and thus obese asthmatics may be more responsive to fish oil. We will determine (in a sub-aim) if there exists an ALOX5 genotype-related response effect with fish oil. This will be the largest clinical trial of omega-3 fatty acid for the treatment of asthma, and the first applying pharmacogenetic/nutrigenetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* age 12-25
* BMI > 25 (age 18-25) or BMI%>85th (age 12-17) (BMI Liberalized)
* Physician diagnosis of persistent asthma
* Lung function responsiveness by bronchodilator reversibility or bronchoprovocation testing

Exclusion Criteria:

* pregnancy
* currently taking LTRA for asthma control
* other serious chronic medical condition
* bleeding diathesis

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2010-07; Primary Completion 2016-10-22 (Actual); Study Completion 2016-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason E. Lang, M.D., Principal Investigator — Duke Children's Hospital and Health Center
Locations (3):
- United States (3):
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Hospital/Dept of Pulmonology, Orlando, Florida
  - University of South Florida, Morsani College of Medicine, Tampa, Florida

REFERENCES:
- [Derived] Lang JE, Mougey EB, Hossain MJ, Livingston F, Balagopal PB, Langdon S, Lima JJ. Fish Oil Supplementation in Overweight/Obese Patients with Uncontrolled Asthma. A Randomized Trial. Ann Am Thorac Soc. 2019 May;16(5):554-562. doi: 10.1513/AnnalsATS.201807-446OC. PMID 30678465

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 were excluded due to medical history and 15 was lost to follow-up during run-in.
Period: Overall Study
Arm/Group | Omega-3 Fatty Acids | Control
Started | 77 | 21
Completed | 68 | 17
Not Completed | 9 | 4
Not completed — Lost to Follow-up | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Fatty Acids | Control | Total
Number analyzed (Participants) | 77 | 21 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (2.2) | 14.6 (2.2) | 14.6 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 11 | 51
  Male | 37 | 10 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 7 | 27
  Not Hispanic or Latino | 57 | 14 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 10 | 50
  White | 30 | 9 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 77 | 21 | 98

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Questionnaire (Juniper)
Description: The ACQ ranges from 0 to 6 (higher values indicate worse asthma control). A score greater than 1.25 in children is considered poor asthma control, and a change of 0.4 or greater is considered clinical meaningful.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Omega-3 Fatty Acids | Control
Number analyzed (Participants) | 77 | 21
score on a scale
  Baseline | 1.13 [0.95 to 1.31] | 1.08 [0.78 to 1.39]
  Change at 3 months | -0.08 [-0.25 to 0.08] | -0.09 [-0.52 to 0.33]
  Change at 6 months | -0.09 [-0.29 to 0.10] | -0.18 [-0.42 to 0.07]
Statistical Analysis 1: Comparison: Omega-3 Fatty Acids vs Control; Test type: Superiority; p = 0.05, ANCOVA

2. Secondary Outcome: N3-to-n6 PUFA Ratio (Granulocytes)
Description: Ratio of total omega-3 to total omega-6 polyunsaturated fatty acids from granulocytes in peripheral blood
Time Frame: Baseline, 3 and 6 months
Population: Blood was not successfully drawn in all children
Measure: Mean (95% Confidence Interval); unit: no units (ratio)
Arm/Group | Omega-3 Fatty Acids | Control
Number analyzed (Participants) | 77 | 21
no units (ratio)
  Baseline: number analyzed (Participants) | 49 | 18
  Baseline | 0.06 [0.03 to 0.08] | 0.10 [0.05 to 0.14]
  3 months: number analyzed (Participants) | 55 | 15
  3 months | 0.19 [0.09 to 0.28] | 0.08 [0.03 to 0.14]
  6 months: number analyzed (Participants) | 41 | 13
  6 months | 0.17 [0.10 to 0.24] | 0.08 [0.02 to 0.14]

3. Secondary Outcome: N3-to-n6 PUFA Ratio (Monocytes)
Description: Ratio of total omega-3 to total omega-6 polyunsaturated fatty acids from monocytes in peripheral blood
Time Frame: Baseline, 3 months, 6 months
Population: blood was not successfully drawn in all children
Measure: Mean (95% Confidence Interval); unit: no units (ratio)
Arm/Group | Omega-3 Fatty Acids | Control
Number analyzed (Participants) | 77 | 21
no units (ratio)
  Baseline: number analyzed (Participants) | 54 | 19
  Baseline | 0.04 [0.03 to 0.05] | 0.08 [0.03 to 0.14]
  3 months: number analyzed (Participants) | 58 | 16
  3 months | 0.11 [0.07 to 0.15] | 0.05 [0.02 to 0.08]
  6 months: number analyzed (Participants) | 44 | 14
  6 months | 0.12 [0.07 to 0.18] | 0.07 [0.03 to 0.11]

4. Secondary Outcome: Asthma Control Test
Description: The asthma control test assesses patient reported symptoms from the prior month and has a range from 5 to 25 with a higher score suggesting better asthma control.
Time Frame: Baseline, 3 months, 6 months
Population: missing data due to drop outs or staff error
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Omega-3 Fatty Acids | Control
Number analyzed (Participants) | 77 | 21
units on a scale
  Baseline: number analyzed (Participants) | 74 | 21
  Baseline | 19.4 [18.5 to 20.2] | 19.9 [18.2 to 21.6]
  3 months: number analyzed (Participants) | 68 | 19
  3 months | 19.5 [18.6 to 20.3] | 20.3 [17.8 to 22.8]
  6 months: number analyzed (Participants) | 67 | 17
  6 months | 20.2 [19.3 to 21.1] | 20.4 [18.0 to 22.7]

5. Secondary Outcome: Urinary Leukotriene-E4
Description: Leukotriene E4 obtained from urine was measured using liquid chromatography tandem mass spectrometry.
Time Frame: Baseline, 3 months, 6 months
Population: missing data resulted from participants lost to follow up or not providing urine samples
Measure: Mean (95% Confidence Interval); unit: pg/mg creatinine
Arm/Group | Omega-3 Fatty Acids | Control
Number analyzed (Participants) | 77 | 21
pg/mg creatinine
  Baseline: number analyzed (Participants) | 67 | 18
  Baseline | 70.1 [59.7 to 80.5] | 84.0 [60.1 to 107.9]
  3 months: number analyzed (Participants) | 62 | 15
  3 months | 78.5 [64.6 to 92.3] | 61.3 [41.4 to 81.1]
  6 months: number analyzed (Participants) | 59 | 12
  6 months | 80.6 [67.9 to 93.3] | 66.5 [43.0 to 90.0]

6. Secondary Outcome: FEV1
Description: Forced expiratory volume in 1 second is a validated spirometry measure.
Time Frame: Baseline, 3 months, 6 months
Population: missing data due to participants lost to follow-up or not being able to provide valid spirometry
Measure: Mean (95% Confidence Interval); unit: percent of predicted
Arm/Group | Omega-3 Fatty Acids | Control
Number analyzed (Participants) | 77 | 21
percent of predicted
  Baseline: number analyzed (Participants) | 74 | 19
  Baseline | 90.2 [86.7 to 93.8] | 90.3 [84.4 to 96.2]
  3 months: number analyzed (Participants) | 69 | 17
  3 months | 91.6 [88.7 to 94.6] | 90.2 [84.1 to 96.3]
  6 months: number analyzed (Participants) | 67 | 15
  6 months | 91.6 [87.4 to 95.8] | 91.7 [85.2 to 98.2]

7. Secondary Outcome: Exacerbations
Description: Exacerbations of asthma were defined by the need for urgent medical care (emergency room or urgent care clinic) or systemic corticosteroids to avoid severe worsening of asthma determined by study physician or local provider
Time Frame: 6 months
Population: all randomized participants
Measure: Number; unit: exacerbations
Arm/Group | Omega-3 Fatty Acids | Control
Number analyzed (Participants) | 77 | 21
exacerbations | 17 | 5

8. Secondary Outcome: Phone Contacts
Description: Phone contact was defined as an urgent or unscheduled phone contact to a medical provider for asthma
Time Frame: 6 months
Population: all randomized participants
Measure: Number; unit: events
Arm/Group | Omega-3 Fatty Acids | Control
Number analyzed (Participants) | 77 | 21
events | 10 | 6

ADVERSE EVENTS:
Time Frame: Over the course of the study post randomization (24 weeks)
Description: Our adverse event and serious adverse event did not differ from the definitions outlined in clinicaltrials.gov.
Arm/Group | Omega-3 Fatty Acids | Control
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/77 | 0/21
Other Adverse Events (participants affected / at risk) | 58/77 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Fatty Acids (N=77) | Control (N=21)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Hospitalized for asthma exacerbation; respiratory distress
vomiting (Gastrointestinal disorders) | 1 (1) | 0 — hematemesis requiring urgent care
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omega-3 Fatty Acids (N=77) | Control (N=21)
Headaches (Nervous system disorders) | 39 | 8 — Painful sensation in any part of the head
Dry Mouth (Immune system disorders) | 14 | 5 — Salivary Glands are not making enough saliva in the mouth
Nausea (Gastrointestinal disorders) | 21 | 4 — Feeling of queasiness or wooziness or need to vomit
Bloating (Gastrointestinal disorders) | 11 | 2 — Intestinal organs are being stretched or distended
Diarrhea (Gastrointestinal disorders) | 11 | 5 — Liquid form of feces discharged from the bowels
Constipation (Gastrointestinal disorders) | 8 | 2 — Difficulty emptying the bowels; harden feces
Flatulence (Gastrointestinal disorders) | 14 | 5 — Accumulation of gas in the stomach
Rash (Skin and subcutaneous tissue disorders) | 15 | 2
URI (Respiratory, thoracic and mediastinal disorders) | 31 | 8 — Infection of the upper respiratory system
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 20 | 8 — Pain and/or inflammation of the throat
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 9 | 1 — Inflamed cavities around the nasal passages

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes